CLINICAL TRIAL: NCT04154735
Title: Autologous Hematopoietic Stem Cell Transplant for Crohn's Disease
Brief Title: Autologous Transplant Targeted Against Crohn's
Acronym: ATTAC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinued by Investigator
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, Division Chief, Immunotherapy and Autoimmune Diseases, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAD.ATTAC.2018
Record Dates: First submitted 2019-03-08; First posted 2019-11-06 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-01

CONDITIONS: Crohn's Disease
Keywords: Autologous Stem Cell Transplantation; Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Crohn Disease | interventions — fludarabine; Cyclophosphamide; Mesna; Alemtuzumab; Granulocyte Colony-Stimulating Factor; Filgrastim; Rifaximin; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Experimental): Hematopoietic Stem Cell Therapy will be performed as follows: Autologous stem cells will be infused after conditioning with fludarabine, cyclophosphamide, mesna, and alemtuzumab. Granulocyte-colony stimulating factor (G-CSF) will be administered post-transplant until engraftment. Rifaximin and tacrolimus will be administered for 6 and 12 months, respectively, beginning one day before the infusion of stem cells.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mesna; Drug: Alemtuzumab; Drug: G-CSF; Drug: Rifaximin; Drug: Tacrolimus

INTERVENTIONS:
Drug: Fludarabine — A chemotherapy medication commonly used in the treatment of leukemia and lymphoma
Drug: Cyclophosphamide — A medication used as chemotherapy and to suppress the immune system
  Other Names: Cytoxan
Drug: Mesna — A medication used in those taking cyclophosphamide or ifosfamide to decrease the risk of bleeding from the bladder
  Other Names: Mesnex
Drug: Alemtuzumab — A protein that kills the immune cells that are thought to be causing Crohn's; it is commonly used in the treatment of leukemia and lymphoma
  Other Names: Lemtrada; Campath
Drug: G-CSF — A glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream
  Other Names: Neupogen; Filgrastim; Granix; Zarxio
Drug: Rifaximin — An antibiotic used to treat irritable bowel syndrome and relapsing C. difficile infection; it inhibits DNA-dependent RNA polymerase
  Other Names: Xifaxan
Drug: Tacrolimus — A medication which suppresses the immune system and inhibits T-lymphocytes; commonly used to lower the risk of organ rejection following transplant
  Other Names: Prograf; Envarsus XR; Stargraf XL

SUMMARY:
This study is a new Phase II trial to assess the toxicity and efficacy of autologous hematopoietic stem cell transplantation (HSCT) utilizing a new non-myeloablative conditioning regimen in patients with high-risk Crohn's disease (CD). The regimen will include low-dose immunosuppressive therapy and a targeted antibiotic for six to twelve months post-HSCT.

DETAILED DESCRIPTION:
The autologous hematopoietic stem cell transplantation (HSCT) in this study utilizes a new non-myeloablative conditioning regimen in patients with high-risk Crohn's disease (CD). The regimen includes two types of chemotherapy (cyclophosphamide and fludarabine) as well as alemtuzumab. The regimen will include low-dose immunosuppressive therapy with tacrolimus (Prograf) for one year post-HSCT in attempt to prevent relapse and improve long-term remission. Patients will also receive rifaximin (Xifaxan) for six months post-HSCT to target abnormal intestinal microbiota that may trigger intestinal inflammation. The ability of these experimental treatments to stop relapses and progression (worsening) of Crohn's disease will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and less than age 50 years at the time of pre-transplant evaluation
2. Ability to give informed consent
3. An established clinical diagnosis of severe Crohn's Disease* that has failed therapy with prednisone or budesonide (Entocort) and either a or b below:

   1. At least two anti-tumor necrosis factor (TNF) drugs (e.g., infliximab (Remicade), adalimumab (Humira), or certolizumab pegol (Cimzia))
   2. One anti-TNF drug as above and either vedolizumab (Entyvio) or ustekinumab (Stelara)

      * Severe Crohn's Disease is defined as a CDAI (see Appendix A) of 250 to 400 or a Craig's Crohn's Severity Index (CCSI, see Appendix B) that is > 17.

Exclusion Criteria:

1. Uncontrolled diabetes mellitus or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment
2. Prior history of malignancy (except localized basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix). Other malignancies for which the patient is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I breast cancer will be considered on an individual basis
3. Positive pregnancy test, inability to pursue effective means of birth control, or failure to willingly accept or comprehend irreversible sterility as a side effect of therapy
4. HIV positive
5. Hepatitis B or C positive
6. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
7. Untreated life-threatening cardiac arrhythmia on EKG or 24-hour holter or history of coronary artery disease or congestive heart failure
8. Left ventricular ejection fraction (LVEF) <50%
9. Forced vital capacity (FVC) <60% of predicted after bronchodilator therapy (if necessary) or diffusing capacity of the lungs for carbon monoxide (DLCO) hemoglobin corrected <60 % predicted
10. Serum creatinine >2 mg/dl
11. 24-hour urine creatinine clearance <90
12. Liver transaminases >2x of normal limits, or bilirubin >2 mg/dl unless due to Crohn's Disease
13. Major hematological abnormalities such as platelet count < 100,000/ul or absolute neutrophil count (ANC) < 1500/ul
14. Failure to collect at least 2 x10^6 cluster of differentiation 34 (CD34+) cells/kg
15. Any active infection
16. Known hypersensitivity to mouse, rabbit, or E. coli derived proteins
17. Short Bowel Syndrome defined as intestinal dysfunction with the presence of significant malabsorption of both macronutrients and micronutrients or when gastrointestinal function is inadequate to maintain nutrient and hydration status without intravenous or enteral supplementation.
18. History of anorexia nervosa (serum albumin ≤ 20 g/L, body mass index ≤ 18)
19. Patients presenting with intestinal perforation or toxic megacolon or a problem that will require urgent surgery. The presence of intestinal stomas, strictures, or fistulae does not exclude the patient from study.
20. Unable or unwilling to stop using and/or smoking tobacco products
21. Abnormal peripheral blood cytogenetics

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Treatment-related mortality | 3 years
  Treatment-related mortality
Overall survival | 3 years
  Survival of participants
Clinical remission | 6 months, 1 year, 2 years, 3 years
  Change of Crohn's Disease Activity Index CDAI ≤ 150, Harvey-Bradshaw Index (HBI) ≤4, may be on immune suppressive drugs
Complete remission | 1 year, 2 years, 3 years
  Change of Clinical, endoscopic, and histologic remission on no immune modulating drugs

SECONDARY OUTCOMES:
Craig's Crohn's Severity Index | 6 months, 1 year, 2 years, 3 years
  Improvement in the severity of Crohn's Disease according to the Craig's Crohn's Severity Index (CDAI)
Endoscopic severity scales | 6 months, 1 year, 2 years, 3 years
  Improvement on the Simple Endoscopic Score for Crohn's Disease (SES-CD)
Histologic remission on colonoscopy with biopsy | 6 months, 1 year, 2 years, 3 years
  No evidence of disease on biopsy
Endoscopic remission | 6 months, 1 year, 2 years, 3 years
  No evidence of disease on colonoscopy
Drug-free clinical remission | 1 year, 2 years, 3 years
  Crohn's Disease Activity Index (CDAI ≤ 150),Harvey Bradshaw Index HBI ≤4, no immune suppressive drugs
Relapse-free survival | 6 months, 1 year, 2 years, 3 years
  Relapse is defined as Crohn's Disease Activity Index CDAI >150, Harvey Bradshaw Index HBI >4, and restarting or increasing immune based medication(s)
Stool markers | 6 months, 1 year, 2 years, 3 years
  Improvement in fecal calprotectin and fecal lactoferrin
Quality of life short form Survey (SF-36) | 6 months, 1 year, 2 years, 3 years
  Improvement in quality of life, measured by 36-Item Short Form Survey (SF-36) The evaluation of the results was done by attributing scores to each question, which were then transformed into a scale ranging from 0 to 100, where 0 corresponds to the worst quality of life and 100 to the best.
Inflammatory Bowel Disease Questionnaire | 6 months, 1 year, 2 years, 3 years
  Improvement on the Inflammatory Bowel Disease Questionnaire (IBDQ) Total IBDQ score ranges from 32 to 224. A higher score indicates better quality of life.
Crohn's Disease Endoscopic Index of Severity (CDEIS) | 6 months, 1 year, 2 years, 3 years
  Improvement on the Crohn's Disease Endoscopic Index of Severity (CDEIS)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No